CLINICAL TRIAL: NCT04957121
Title: Comparison of Anesthesia Beginning at On-hours Versus Off-hours on Outcomes in Patients Undergoing Hip Surgery
Brief Title: Comparison of On-hours Versus Off-hours Anesthesia of Hip Surgery
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, Deputy Director of Anesthesiology Department of Tongji Hospital Affiliated to Huazhong University of Science and Technology, Huazhong University of Science and Technology
Other Study IDs: TJ-IRB20210305
Record Dates: First submitted 2021-06-21; First posted 2021-07-12 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Off-hours Anesthesia
Keywords: off-hours; hip surgery; perioperative care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- on-hours: Hip surgeries with the start time of anesthesia between 8:00 and 17:59 were coded as "on-hours".
  Interventions: Other: on-hours
- off-hours: Hip surgeries with anesthesia beginning between 18:00 and 7:59 were coded as "off-hours". Besides, taking the long duration of hip surgery into account, if the anesthesia began before 18:00 but ended after 20:00, it was also defined as "off-hours".
  Interventions: Other: off-hours

INTERVENTIONS:
Other: on-hours — If the begin time of anesthesia was between 8:00 to 17:59, it was defined as "on-hours".
  Groups: on-hours
Other: off-hours — If the start time of anesthesia was between 18:00 to 7:59 or the end time of anesthesia was later than 20:00, it was defined as "off-hours".
  Groups: off-hours

SUMMARY:
To explore the impact of the begin time of anesthesia on in-hospital mortality and early prognosis of patients undergoing hip surgery.

DETAILED DESCRIPTION:
The patients undergoing hip surgery between were divided into the on-hours group or the off-hours group depending on the begin time of anesthesia in this retrospective cohort study. In-hospital mortality and early prognosis were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* All patients who had hip surgery between January 1, 2015, and December 31, 2020 in Tongji Hospital.

Exclusion Criteria:

* under 18 years old
* had incomplete perioperative data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had hip surgery during on-hours or off-hours.
Sampling Method: Non-Probability Sample
Enrollment: 1843 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2021-08-08 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
in-hospital mortality | up to 7 months
  the mortality during hospitalization

SECONDARY OUTCOMES:
postoperative LOS | up to 4 months postoperatively
  postoperative hospital length of stay
total LOS | up to 7 months
  total hospital length of stay
ICU admission | within 3 days postoperatively
  the ratio of ICU admission
postoperative complications | within 3 days postoperatively
  including renal dysfunction, anemia, hypotension, deep vein thrombosis, arrhythmia, coronary artery disease or heart failure, pulmonary infection, electrolyte disturbance, hyoxemia and delirium
intraoperative fluid management | intraoperative
  including blood loss, urine volume, concentrated red blood cells, fresh frozen plasma, equilibrium liquid and colloidal solution
intraoperative sufentanil | intraoperative
  the dosage of intraoperative sufentanil
using vasoactive drugs | intraoperative
  whether using vasoactive drugs or not intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Wei Mei, Principal Investigator — Tongji Hospital
Locations (1):
- Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No